CLINICAL TRIAL: NCT01587742
Title: IMI PROTECT (Work Package 2): Calcium Channel Blocker Treatments and Cancer Risk
Brief Title: IMI PROTECT (Work Package 2): Calcium Channel Blockers and Cancer
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115736; WEUKBRE5558 (Other: GSK)
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension
Keywords: Calcium channel blockers; cancer
MeSH Terms: conditions — Hypertension; Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Patients with a diagnosis of any cancer type: All patients of the study population with a diagnosis of any cancer type based on Read codes and ICD-10 codes
  Interventions: Drug: CCB use
- Patients with a diagnosis of breast cancer: All patients of the study population with a diagnosis of breast cancer based on Read codes and ICD-10 codes
  Interventions: Drug: CCB use
- Patients with a diagnosis of prostate cancer: All patients of the study population with a diagnosis of prostate cancer based on Read codes and ICD-10 codes
  Interventions: Drug: CCB use
- Patients with a diagnosis of colon cancer: All patients of the study population with a diagnosis of colon cancer based on Read codes and ICD-10 codes
  Interventions: Drug: CCB use
- Patients without a diagnosis of any cancer type: All patients of the study population without a diagnosis of any cancer type
  Interventions: Drug: CCB use

INTERVENTIONS:
Drug: CCB use — Prescription of CCB during the study period between January 1, 1996 to December 31, 2009. The CCBs administered to the patients include isradipine and lacidipine.

SUMMARY:
The studies described in this protocol are all performed within the framework of PROTECT (Pharmacoepidemiological Research on Outcomes of Therapeutics by a European ConsorTium) Workpackage 2 (WP2) and Workgroup 1. The primary aim of these studies is to develop, test and disseminate methodological standards for the design, conduct and analysis of Pharmacoepidemiological (PE) studies applicable to different safety issues and using different data sources. To achieve this, results from PE studies on 5 key adverse events (AEs) performed in different databases will be evaluated. Therefore, emphasis will be on the methodological aspects of the studies in this protocol and not on the clinical consequences of the association under investigation. The standards to develop will contribute to decreasing the discrepancies in results from different studies in the future and increase the usefulness and reliability of these studies for benefit-risk assessment in the EU.

Within WP2, five possible adverse event - drug pairs have been selected for analyses; one of these includes the possible role of calcium channel blockers (CCBs) in the risk of cancer. Analyses will address the hypothesis that CCBs modify the risk of cancer (all forms of cancer combined and various groups of cancers).

This hypothesis will be investigated using two sources of data: the UK General Practice Research Database (GPRD) and the Danish national databases. Investigations in the UK may also use The Health Improvement Network (THIN).

The primary objective of the study is to investigate the possible association between use of CCBs and risk of all forms of cancer combined, among adult patients (18 to 79 years of age during the study period, January 1, 1996 to December 31, 2009). The study will be conducted using three databases with different study designs (descriptive, cohort, population based cohort study and nested case-control) across different databases (GPRD, THIN, Danish databases) and to compare the results between databases, across designs to evaluate the impact of design/database/population differences on the outcome of the studied association.

Secondary objectives are to investigate the potential association between use of CCBs and risk of all forms of breast cancer in women; all forms of prostate cancer; and all forms of colon cancer using the same age groups and databases).

DETAILED DESCRIPTION:
Conducting studies on the possible association between CCBs and cancer using a pharmaco-epidemiological approach based on data collected in existing databases and cancer registries is challenging. The challenge lies in working within the limitations of the available data (in terms of quality and completeness) and simultaneously maximizing the value of the available data through thoughtful study design and statistical analysis.

CCBs represent a chemically and pharmacologically diverse group of agents that are widely used for the treatment of hypertension and angina. It has been proposed that CCBs may interfere with apoptosis, leading to an increased potential for abnormal cell proliferation and tumor growth. The underlying biological mechanism for this effect is thought to be linked to the role of transmembrane Ca2+. This hypothesis has been critically reviewed and results have shown that the action of CCBs on apoptosis are complex with both increases and decreases in intracellular Ca2+ linked to this form of programmed cell death (2). CCBs have also been shown to inhibit apoptosis in certain non-transformed cell lines but promote apoptosis in other non-transformed and transformed cell lines. The results from non-human genotoxicity studies have shown no link between CCB use and tumor development

Epidemiologic studies have also provided inconsistent results. While only a few follow-up analyses reported an increased risk for all cancer or breast cancer, further observational studies have so far provided no evidence to support the hypothesis that long-term use of CCBs might be carcinogenic. As a whole, these studies have been limited by lack of statistical power and/or inadequate methods for defining the exposure window of antihypertensive treatment in relation to the index date (cancer outcome), making the establishment of a causal relationship between CCBs use and risk of cancer problematical. Studies often assumed a relatively short period of CCB use (usually between 2 months and 1 year) before entering the study as users. In other cases, information on the use of CCBs was only available at study entry or during follow-up. Overall, most studies were limited by follow-up periods that could be considered too brief to measure a carcinogenic effect. The vast majority of studies collected information from electronic medical or administrative databases.

The current study aims to learn from the experience, strengths and limitations of previous research to present a best-practice approach to addressing the hypothesis in question. Combined with the objectives of the PROTECT program, we hope that this study will help to provide a framework for guiding methodological choices in future research and contribute to increasing the usefulness and reliability of pharmacoepidemiological studies for benefit-risk assessment and decision making.

ELIGIBILITY:
Inclusion Criteria:

* First time users or non-users of a CCB from January 1, 1996 to December 31, 2009
* Patients aged 18 to 79 years

Exclusion Criteria:

* Patients with any cancer recorded in the GPRD or the Danish database prior to cohort entry
* Patients aged less than 18 years or more than 79 years

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of CCB first-time users and non-users from January 1, 1996 to December 31, 2009, aged 18 to 79 years enrolled in the GPRD, THIN or Danish National database
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in incidence of primary cancer (all forms) cases, defined by Read codes in GPRD/THIN and ICD-10 codes in the Danish data | During Jan 1, 1996 to Dec 31, 2009 , cancer outcomes will be assessed as those occurring six months - 1 year, 1-4 years and more than 5 years following initiation of CCB therapy

SECONDARY OUTCOMES:
Change in incidence of breast cancer cases in women only defined by Read codes in GPRD/THIN and ICD-10 codes in the Danish data | During Jan 1, 1996 to Dec 31, 2009, cancer outcomes will be assessed as those occurring six months - 1 year, 1-4 years and more than 5 years following initiation of CCB therapy
Change in incidence of prostate cancer cases only, defined by Read codes in GPRD/THIN and ICD-10 codes in the Danish data | During Jan 1, 1996 to Dec 31, 2009, cancer outcomes will be assessed as those occurring six months - 1 year, 1-4 years and more than 5 years following initiation of CCB therapy
Change in incidence of colon cancer cases only, defined by Read codes in GPRD/THIN and ICD-10 codes in the Danish data | During Jan 1, 1996 to Dec 31, 2009, cancer outcomes will be assessed as those occurring six months - 1 year, 1-4 years and more than 5 years following initiation of CCB therapy

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline